CLINICAL TRIAL: NCT06997952
Title: Impact of Febuxostat on Disease Progression and Carotid Intima-Media Thickness in Patients With Chronic Kidney Disease
Brief Title: Febuxostat Effect on Chronic Kidney Disease Progression And Carotid Intima-Media Thickness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS268/2024
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Carotid Intima- Media Thickness
MeSH Terms: interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Active Comparator): Received febuxostat daily for 12 weeks in addition to their standard treatment. The prescribed dosage was 40 mg taken once daily, self-administered by the patients.
  Interventions: Drug: Febuxostat 40 mg
- Control (No Intervention): continued with their standard treatment alone

INTERVENTIONS:
Drug: Febuxostat 40 mg — Febuxostat will be given daily for 12 weeks The prescribed dosage was 40 mg taken once daily, self-administered by the patients in addition to their standard treatment.
  Arms: Case

SUMMARY:
This study aimed to evaluate the impact of febuxostat on both carotid intima-media thickness and disease progression in individuals with chronic kidney disease

DETAILED DESCRIPTION:
For all participants, comprehensive data collection was performed, encompassing detailed medical histories including patients' clinical and demographic characteristics (age, gender, BMI, associated comorbidities as HTN, and DM, etiology of CKD.) Laboratory investigations were conducted at baseline and after a three-month follow-up period. These investigations included: serum uric acid., creatinine, blood urea nitrogen, calcium, phosphorus., albumin., magnesium, intact parathyroid hormone (iPTH), lipid profile (cholesterol, triglycerides, LDL, HDL), urine protein to creatinine ratio. Radiological investigations: Carotid artery duplex (medial wall thickness) was also conducted at baseline and after a three-month follow-up period. Thickening of the artery wall is a hallmark of atherosclerosis and vascular calcification.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* CKD stages III to IV
* Asymptomatic hyper uricemia
* Stable dose of all medications including ACEIs or ARBs for blood pressure control at least three months before enrolling

Exclusion Criteria:

* Comprised active infections.
* Acute kidney injury.
* Active and advanced malignancy.
* History of hypersensitivity to febuxostat.
* Women who are taking oral contraceptives, pregnant or lactating
* Patients with established cardiovascular disease.
* Patients with liver disease.
* Patients receiving mercaptopurine, theophylline and azathioprine.
* Patients on steroids or other immunosuppressive treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
slowing CKD progression | 3 month
  improvement of eGFR and proteinuria after 12 weeks of administration of febuxostat (slowing CKD progression), compared with that of the control group.

SECONDARY OUTCOMES:
improvement of carotid intima-media thickness | 3 month
  improvement of carotid intima-media thickness after after 12 weeks of administration of febuxostat ,compared with that of the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: May 24, 2024, to August 24, 2024